CLINICAL TRIAL: NCT06807437
Title: A Randomized Phase III Blinded Trial of Lanreotide for the Prevention of Postoperative Pancreatic Fistula
Brief Title: Lanreotide Versus Placebo Before Surgery to Prevent a Surgical Complication Called a Pancreatic Fistula
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S2408; NCI-2024-08361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2408 (Other: SWOG); SWOG-S2408 (Other: DCP); S2408 (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Carcinoma; Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Specimen Handling; lanreotide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant, surgeon, and the clinical care team are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (lanreotide, distal pancreatectomy) (Experimental): Patients receive lanreotide SC over 20 seconds and within 36 hours of planned distal pancreatectomy. Patients also undergo blood sample collection immediately prior to surgery and on post-operative days 1 and 3. Additionally, patients may undergo collection of pancreas fluid on post-operative days 1 and 3.
  Interventions: Procedure: Biospecimen Collection; Procedure: Distal Pancreatectomy; Drug: Lanreotide; Other: Questionnaire Administration
- Arm II (saline placebo, distal pancreatectomy) (Placebo Comparator): Patients receive saline placebo SC over 20 seconds and within 36 hours of planned distal pancreatectomy. Patients also undergo blood sample collection immediately prior to surgery and post-operatively on days 1 and 3. Additionally, patients may undergo collection of pancreas fluid on post-operative days 1 and 3.
  Interventions: Procedure: Biospecimen Collection; Procedure: Distal Pancreatectomy; Other: Questionnaire Administration; Other: Saline

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample and pancreas fluid collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Distal Pancreatectomy — Undergo distal pancreatectomy
Drug: Lanreotide — Given SC
  Other Names: Angiopeptin; BIM-23014; DC 13116; Dermopeptin; Ipstyl; Somatulina; Somatuline
  Arms: Arm I (lanreotide, distal pancreatectomy)
Other: Questionnaire Administration — Ancillary studies
Other: Saline — Given SC
  Other Names: ISOTONIC SODIUM CHLORIDE SOLUTION; Normal Saline; Sodium Chloride 0.9%
  Arms: Arm II (saline placebo, distal pancreatectomy)

SUMMARY:
This phase III trial compares the effect of using lanreotide before surgery to surgery alone in preventing pancreatic fistulas in patients with pancreatic cancer or a pancreatic lesion that could become cancerous. Lanreotide, a type of somatostatin analog similar to somatostatin (a hormone made by the body), and is used to treat certain types of gastroenteropancreatic neuroendocrine tumors, and carcinoid syndrome. It may help stop the body from making extra amounts of certain hormones, including growth hormone, insulin, glucagon, and hormones that affect digestion. It may also help keep certain types of tumor cells from growing. Patients with pancreatic cancer or pancreatic lesions may undergo surgery to remove parts of the pancreas, also called a distal pancreatectomy. Patients may experience complications after surgery, including pancreatic fistulas. A pancreatic fistula occurs when there is a small leak from the pancreas, causing fluids to collect. This can often lead to infection and other problems. Giving lanreotide before undergoing distal pancreatectomy may be more effective than surgery alone in preventing the development of a pancreatic fistula in patients with pancreatic cancer or a pancreatic lesion that could become cancerous.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the incidence of postoperative pancreatic fistula (POPF) occurring within 60 days after surgery in participants randomized to receive preoperative lanreotide versus placebo prior to undergoing distal pancreatectomy for biopsy-proven or suspected neoplasm.

SECONDARY OBJECTIVES:

I. To compare the incidence of International Study Group of Pancreatic Surgery (ISGPS)-defined biochemical leak occurring within 60 days after surgery in participants randomized to receive preoperative lanreotide versus placebo in the subset of participants with a drain placed.

II. To compare the number of postoperative days in the hospital within 60 days after surgery in participants randomized to receive preoperative lanreotide versus placebo.

III. To compare change from baseline in cancer-specific quality of life at 14 and 60 days after surgery, as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30-(C30), in participants randomized to receive preoperative lanreotide versus placebo.

ADDITIONAL OBJECTIVES:

I. To compare change from baseline in pancreatic cancer-specific quality of life and overall health-related quality of life at 14 and 60 days after surgery, as measured by the EORTC QLQ- Pancreatic Cancer 26 (PAN26) and European Quality of Life Five Dimension Five Level (EQ-5D-5L), in participants randomized to receive preoperative lanreotide versus placebo.

II. To compare the proportions of participants with common postoperative sequelae associated with POPF, including ISGPS delayed gastric emptying and ISGPS post pancreatectomy hemorrhage (grades B/C) occurring within 60 days after surgery, in participants randomized to receive preoperative lanreotide versus placebo.

III. To compare time from surgery to initiation of adjuvant chemotherapy among participants with pancreatic ductal adenocarcinoma and planned adjuvant chemotherapy randomized to receive preoperative lanreotide versus placebo.

BANKING OBJECTIVE:

I. To bank blood, pancreas fluid, and tissue specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive lanreotide subcutaneously (SC) over 20 seconds and within 36 hours of planned distal pancreatectomy. Patients also undergo blood sample collection immediately prior to surgery and on post-operative days 1 and 3. Additionally, patients may undergo collection of pancreas fluid on post-operative days 1 and 3.

ARM II: Patients receive saline placebo SC over 20 seconds and within 36 hours of planned distal pancreatectomy. Patients also undergo blood sample collection immediately prior to surgery and post-operatively on days 1 and 3. Additionally, patients may undergo collection of pancreas fluid on post-operative days 1 and 3.

After completion of study treatment, patients are followed up at 4, 8 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or radiographically confirmed diagnosis of pancreatic cancer or a pancreatic lesion with malignant potential
* Participants must have an elective distal pancreatectomy planned to occur within 60 days after registration/randomization date
* Participants must not have a known history of a prior diagnosis of malabsorption syndrome
* Participants must not have been treated with any somatostatin analogue within 180 days prior to registration/randomization
* Participants must not have been treated with radiation therapy for their pancreas malignancy at any time prior to registration/randomization
* Participants must not have been treated with peptide receptor radionuclide therapy (PRRT) at any time prior to registration/randomization
* Participants must be ≥ 18 years old
* Participants must have a complete documented medical history and physical exam within 28 days prior to registration/randomization
* Participants must have a creatinine ≤ the institutional upper limit of normal (IULN) OR a measured OR calculated creatinine clearance ≥ 50 mL/min using the following Cockcroft -Gault formula within 60 days prior to registration/randomization
* Participants must complete a pre-registration screening to identify any of the medications below, allowing the study team and treating physician to develop a monitoring plan as needed. Participants taking medications with known interactions with lanreotide may remain eligible if appropriate monitoring and management are in place. These medications include:

  * Diabetes medications (insulin or oral hypoglycemics): Blood sugar will be monitored, and medication dose adjustments made as needed
  * Cyclosporine: Dosage adjustments may be required to maintain therapeutic levels
  * Bromocriptine: Dose adjustments may be considered to account for absorption changes
  * Heart medications (e.g., beta blockers): Heart rate will be monitored, and medication doses adjusted if necessary
  * CYP3A4-metabolized medications: Dose adjustments may be considered to avoid increased exposure
* In the opinion of the treating surgeon, based on preoperative data, the participant must not require a modified Appleby-type procedure (distal pancreatectomy with celiac axis resection) or multivisceral resection (e.g., stomach, colon, etc.) at the time of distal pancreatectomy

  * NOTE: planned removal of the gallbladder or spleen at the time of distal pancreatectomy is not considered multivisceral resection and is permissible
* In the opinion of the treating surgeon, based on preoperative data, the participant must not require a tumor enucleation
* Participants must not have moderate to severe hepatic impairment as defined by liver enzyme elevation more than 5 times the institutional upper limit of normal (either aspartate aminotransferase [AST] > 190 U/L or alanine aminotransferase [ALT] > 320 U/L) within 60 days prior to registration/randomization. Transient elevation at the time of screening that resolves prior to study enrollment is acceptable
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped)
* Individuals who are of reproductive potential must have agreed to use an effective contraceptive method during the whole period of the study and for three months after the study drug administration, with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must be offered the opportunity to participate in specimen banking
* Participants who can complete EORTC QLQ-C30, EORTC QLQ-PAN26, and EQ-5D-5L forms in English or Spanish, must be offered the opportunity to participate in the quality-of-life study
* NOTE: As a part of the OPEN registration process, the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
* For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pancreatic fistula (POPF) | Up to 60 days after distal pancreatectomy
  POPF will be assessed using the 2016 International Study Group for Pancreas Surgery (ISGPS). Incidence rates of POPF in each treatment arm will be described, and treatment arm differences assessed via logistic regression model with adjustment for stratification factor.

SECONDARY OUTCOMES:
Incidence of biochemical leak (BL) | Up to 60 days after distal pancreatectomy
  BL will be defined by the ISGPS as a peritoneal drain amylase greater than three times the upper limit of the institutional normal serum amylase without an effect on clinical management or duration of hospital stay. BL will only be measured in those who had a peritoneal drain placed. Treatment arm differences will be assessed via logistic regression model with adjustment for stratification factor.
Number of post-operation hospital days | From the time of surgery up to 60 days after distal pancreatectomy
  Mean hospital length of stay will be compared according to treatment arm via linear regression model with adjustment for stratification factor.
Change in overall quality of life (QOL) | At baseline and at 14 and 60 days after surgery
  Assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ) Core 30 (C30). Treatment arm differences in EORTC QLQ-C30 changes will be assessed by repeated measures linear regression model as a function of randomization assignment, baseline score, stratification factor, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures.

OTHER OUTCOMES:
Changes in pancreatic specific QOL | At baseline and up to 60 days after distal pancreatectomy
  Will be assessed using EORTC QLQ- Pancreatic Cancer 26. Treatment arm differences in changes from baseline will be assessed by repeated measures linear regression model as a function of randomization assignment, baseline score, stratification factor, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures.
Change in health-related QOL | At baseline and up to 60 days after distal pancreatectomy
  Will be assessed using the European Quality of Life Five Dimension Five Level scale. Treatment arm differences in changes from baseline will be assessed by repeated measures linear regression model as a function of randomization assignment, baseline score, stratification factor, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures.
Delayed gastric emptying (DGE) | Up to 60 days after distal pancreatectomy
  DGE will be defined by the ISGPS as reinsertion or persistence of a nasogastric tube after postoperative day (POD) 3 or inability to tolerate solid oral intake by POD 7. Treatment arm differences in the proportion of participants with DGE will be assessed via logistic regression model with adjustment for stratification factor.
Incidence of grades B/C post-pancreatectomy hemorrhage (PPH) | Up to 60 days after distal pancreatectomy
  PPH will be defined by the ISGPS as postoperative intra- or extra-luminal hemorrhage requiring transfusion of fluid or blood, intensive care unit transfer, therapeutic endoscopy, endovascular embolization, or reoperation. Treatment arm differences in the proportion of participants with PPH will be assessed via logistic regression model with adjustment for stratification factor.
Time to initiation of adjuvant chemotherapy | From date of surgery to date of first dose of adjuvant chemotherapy up to 60 days after distal pancreatectomy
  Distributions of time from surgery to initiation of adjuvant chemotherapy, among participants with planned adjuvant chemotherapy, in each arm will be estimated via cumulative incidence and compared using the stratified log-rank test.
Incidence of nausea and vomiting | Up to 60 days after distal pancreatectomy
  Proportions of participants with any nausea/vomiting will be compared between treatment arms via Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Sham, Principal Investigator — SWOG Cancer Research Network
Locations (93):
- United States (93):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Saint Joseph's Crosslake Clinic, Crosslake, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Essentia Health - Saint Joseph's Pequot Lakes Clinic, Pequot Lakes, Minnesota
  - Essentia Health - Saint Joseph's Pine River Clinic, Pine River, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health - Saint Joseph's Staples Clinic, Staples, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - State University of New York Upstate Medical University, Syracuse, New York
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Tamarack Health Hayward Medical Center, Hayward, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin